CLINICAL TRIAL: NCT01413308
Title: Long-term Effects on Pulmonary Function in Post- Fontan Operation
Brief Title: Pulmonary Functions Test in Patients After Fontan Operation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Asaad Khoury MD, Rambam health care campus
Other Study IDs: 0148CTIL
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Fontan Operation
Keywords: Fontan; lung function test; nitric oxide production; NYHA class 1-2 without acute or chronic specified lung disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Developed in the early 1970s, Fontan Operation has provided palliative care for patients with single ventricle physiology. Single ventricle is a rare subclass of the atrioventricular (AV) alignment abnormalities double inlet and common inlet ventricles (and rarely, straddling tricuspid valve), in which there is only one ventricular sinus [1]. Most patients present with symptoms of congestion , low cardiac output, and deep cyanosis immedietly after birth. Untreated, these heart anomalies are highly lethal. Neonatal heart transplantation is implacable because of shortage of donors. Fontan operation is a three staged palliative procedure: the single ventricle pumping blood to the systemic circulation , while blood flows laminarly to the lungs through direct anastomosis of the superior and inferior vena cavae (total cavo pulmonary connections), inevitably by-passing the right heart .

This procedure has been shown to immediately correct the mixed venous blood dysfunction, providing treatment for the prominent signs of cyanosis.

Along with its beneficial outcomes, Fontan circulation patients have been documented to have a variety of post-operative late complications. Of most substantial, increased systemic vascular resistance (mean of 10-15 mmHg higher) [2], systolic dysfunction as a result of decreased preload and increase afterload [3], and atrial arrhythmias [4].

With the advent of bypassing right-heart circulation with Fontan operation, the pulmonary vascular bed is exposed to a new atmosphere of blood flow. Instead of physiological pulsatile flow in normal circulation, the pulmonary vasculature is receiving slow velocity, laminar flow [5]. Patients post-Fontan operations have been documented to have restrictive-type pulmonary function, but still yet to be correlated with Fontan circulation or as a possible result of prior lung tissue injury from the pre/intra-operation high volume blood flow. Regardless, Fontan patients are described to have decreased pulmonary function.

The purpose of this research effort is to document and analyze the pulmonary function of those patients post-Fontan operation. It is still unclear as to what the long-term effects of Fontan operation are towards the pulmonary vascular bed, leaving us questions about the effects on lung capacities, ventilation-perfusion efficiency, and oxygen saturation.

DETAILED DESCRIPTION:
Generation of Data:

1. Spirometry-Spirometry will be performed in accordance with ATS/ERS (American Thoracic Society/ European Respiratory Society) Task Force using a KoKo spirometer (KoKo system, PDS Inc., Ferraris Cardiopulmonary System Group; Louisville, CO, USA). Each maneuver will be repeated for at least three technically acceptable FEFV curves; the best results were used for analysis. [6]
2. Whole Body Plethysmography- FRCpleth will be measured in a commercial, whole body ZAN500 constant volume body plethysmograph (ZAN-Messgeraete GmbH, Germany); the surrounded glassed cabin of 980 L includes a chair with adjustable height, all meeting the ATS/ERS recommendations for plethysmography measurements [7,8]. The flow, volume, cabin pressure, and mouth pressures are automatically calibrated. BTPS conditions for lung volumes are automatically corrected. According to the manufacturer, environmental interference is automatically reduced by a numeric-drift-compensation, enabling quick stable signals for immediate testing.
3. MCT - Methacholine challenge tests will be performed in a designated room at the Pediatric Pulmonary Unit, Meyer Children's Hospital, Haifa, Israel. MCT was performed with double doses of fresh methacholine solutions in saline. Solutions were driven by KoKo-PDS dosimeter via mouthpiece. The MCT will end when FEV1 dropped by more 20% from baseline FEV1 values or when a methacholine concentration of 16 mg/ml was reached. The exact PC20 value will be then calculated by the program according to the log-transformed formula, as described in the guidelines for methacholine.[9] Airway hyper-reactivity was defined as PC20 <8 mg/ml. Oxygen saturation and heart rate were monitored by pulse oximetry (Nonin Wrist Ox 3100, Nonin Medical, Inc., Plymouth, MN, USA).
4. FENO: Measurement of FENO will be performed by portable electrochemical analyzer NIOX MINO (Aerocrine AB, Smidesvägen, Sweden),[10] and according to ATS recommendations . The measurement procedure includes a deep inhalation to total lung capacity followed by exhalation for 10 seconds at a mouth flow rate of 50 mL/sec and a pressure of 10 cmH2O.[11] Analysis of Data: Subjects of study will be patients post-Fontan operation over the age of 6 years in order to fulfill the cooperation requirement necessary to obtain data. Patients should be in general good health without any ongoing acute pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Fontan patient NYHA 1-2
* Age - 10-99

Exclusion Criteria:

* Pregnant woman
* Acute pulmonary disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total number of 15 Fontan patients , aged 10 years and older , with 1-2 NYHA class functional capacity. All will have total pulmonary function tests according to recognized pulmonary protocols. Results will be normalized to age-dependent pulmonogram. Exclusion criteria includes patients with acute pulmonary illness.
  Generation of Data:
  1. Spirometry-Spirometry will be performed in accordance with ATS/ERS (American Thoracic Society/ European Respiratory Society) Task Force
  2. Whole Body Plethysmography- FRCpleth will be measured
  3. MCT - Methacholine challenge tests will be performed
  4. FENO: Measurement of FENO will be performed by portable electrochemical analyzer NIOX MINO (Aerocrine AB, Smidesvägen, Sweden),[10] and according to ATS recommendations .
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Asaad khoury, MD, Principal Investigator — Rambam Health Care Campus